CLINICAL TRIAL: NCT06079359
Title: A Phase 3, Randomized, Double-blinded, Placebo-controlled, Multicenter Study to Evaluate Efficacy and Safety of ALXN1850 Versus Placebo Administered Subcutaneously in Pediatric (2 to < 12 Years of Age) Participants With Hypophosphatasia Who Have Not Received Previous Treatment With Asfotase Alfa
Brief Title: Phase 3 Study of ALXN1850 in Treatment-Naïve Pediatric Participants With HPP
Acronym: MULBERRY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8590C00003; ALXN1850-HPP-305 (Other: Alexion Pharmaceuticals, Inc.)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hypophosphatasia
Keywords: Hypophosphatasia; HPP; ALXN1850
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALXN1850 (Experimental): Starting at Day 1 of the Randomized Evaluation Period, the ALXN1850 group will receive bodyweight dependent doses of either 20mg, 35mg or 50mg of ALXN1850 once every 2 weeks (q2w) via SC injection, for 24 weeks. Participants will enter the OLE Period and continue q2w dosing with ALXN1850 for up to 132 weeks.
  Interventions: Drug: ALXN1850; Drug: Placebo
- Placebo (Placebo Comparator): Starting at Day 1 during the Randomized Evaluation Period, participants will receive placebo q2w for a total of 24 weeks. Participants will enter the OLE Period and continue q2w dosing with ALXN1850 for up to 132 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALXN1850 — Participants will receive a ALXN1850 via subcutaneous (SC) injection.
  Arms: ALXN1850
Drug: Placebo — Participants will receive placebo via SC injection.

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of ALXN1850 versus placebo on radiographic outcomes in pediatric participants with HPP who have not previously been treated with asfotase alfa.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HPP documented in the medical records, and the following criteria fulfilled without other probable cause than HPP:

  1. Presence of HPP-related rickets on skeletal X-rays during the Screening Period, with a minimum Rickets Severity Score (RSS) of 1.0 AND
  2. Serum ALP activity below the age- and sex-adjusted normal range during the Screening Period as measured by the Central Laboratory OR 2 documented serum ALP activity results, at least 15 days apart, below the age- and sex-adjusted local laboratory normal range during the 24 months before the Day 1 Visit. Note: Local laboratories need to be Clinical Laboratory Improvement Amendments (CLIA) or ISO 15189 certified, or have other local equivalent laboratory certification with Alexion's approval.
* Must meet 1 of the following criteria:

  1. Documented ALPL gene variant (pathogenic, likely pathogenic, or variant of unknown significance) from a CLIA certified laboratory (Section 8.7)
  2. Plasma PLP above the upper limit of normal (ULN) during the Screening Period (central or local laboratory results allowed per local regulations)
* Tanner stage 2 or less during the Screening Period

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, neurological disorders, or any other disorders that are capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data as determined by the Investigator
* Diagnosis of primary or secondary hyperparathyroidism
* Hypoparathyroidism, unless secondary to HPP
* Any new fracture within 12 weeks before Day 1 (excluding pseudofractures)
* Planned surgical intervention which may impact the results of study assessments (in the opinion of the Investigator) during the Randomized Evaluation Period
* History of allergy or hypersensitivity to any ingredient contained in ALXN1850 or the placebo comparator

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2028-08-24 (Estimated)

PRIMARY OUTCOMES:
Radiographic Global Impression of Change (RGI-C) Score at the end of the Randomized Evaluation Period (Day 169) | Day 169

SECONDARY OUTCOMES:
Change from Baseline in Rickets Severity Score (RSS) at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
Change from Baseline in 6-Minute Walk Test (6MWT) at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
Change from Baseline in Percent Predicted 6MWT at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
Change from Baseline in Bruininks Oseretsky Test of Motor Proficiency, Second Edition (BOT2) Score at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
Change from Baseline in Peabody Developmental Motor Scales, Third Edition (PDMS-3) Score at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
RGI-C Responder at the end of the Randomized Evaluation Period (Day 169) | Day 169

CONTACTS AND LOCATIONS:
Locations (31):
- United States (3):
  - Research Site, Baltimore, Maryland
  - Research Site, Kansas City, Missouri
  - Research Site, Durham, North Carolina
- Australia (2):
  - Research Site, Nedlands
  - Research Site, Parkville
- Research Site, Brussels, Belgium
- Brazil (5):
  - Research Site, Brasília
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Salvador
  - Research Site, São Paulo
- Canada (2):
  - Research Site, Calgary, Alberta
  - Research Site, Winnepeg, Manitoba
- China (4):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Shanghai
  - Research Site, Shenzhen
- Research Site, Helsinki, Finland
- Research Site, Ashkelon, Israel
- Research Site, Chihuahua City, Mexico
- Research Site, Lodz, Poland
- Research Site, Bucharest, Romania
- Spain (2):
  - Research Site, Madrid
  - Research Site, Vitoria-Gasteiz
- Research Site, Stockholm, Sweden
- Research Site, Taipei, Taiwan
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Erzurum
  - Research Site, Istanbul
- Research Site, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR